CLINICAL TRIAL: NCT01530100
Title: Lower Laser Therapy in Orthognathics Surgery - Double Blind Study.
Brief Title: Lower Laser Therapy in Orthognathics Surgery
Status: Completed | Type: Observational
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Giovanni Gasperini, master, Universidade Federal de Goias
Other Study IDs: LLTOS
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2012-02

CONDITIONS: Dentofacial Deformity
Keywords: Edema; Pain; Lower laser therapy; orthognathics surgery
MeSH Terms: conditions — Dentofacial Deformities; Edema; Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will examine the use of lower laser therapy to reduce edema and pain in orthognathics surgery.

ELIGIBILITY:
Inclusion Criteria:

* Dentofacial deformity
* Healthy
* Mandibular surgery
* no medication use

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
edema, pain and neurosensory disturbancy | 2 months
  edema, pain and neurosensory disturbancy, response to lasr therapy

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Gasperini, master, Principal Investigator — UFG

REFERENCES:
- [Derived] Gasperini G, Rodrigues de Siqueira IC, Rezende Costa L. Does low-level laser therapy decrease swelling and pain resulting from orthognathic surgery? Int J Oral Maxillofac Surg. 2014 Jul;43(7):868-73. doi: 10.1016/j.ijom.2014.02.015. Epub 2014 Mar 25. PMID 24679851
- [Derived] Gasperini G, de Siqueira IC, Costa LR. Lower-level laser therapy improves neurosensory disorders resulting from bilateral mandibular sagittal split osteotomy: a randomized crossover clinical trial. J Craniomaxillofac Surg. 2014 Jul;42(5):e130-3. doi: 10.1016/j.jcms.2013.07.009. Epub 2013 Sep 4. PMID 24011464